CLINICAL TRIAL: NCT01270516
Title: Effect of EPA and HMB on Diaphragm and Limb Muscle Strength in Mechanically Ventilated Patients
Brief Title: Effect of EPA and HMB on Strength in ICU Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerald Supinski (Other)
Responsible Party: Sponsor-Investigator, Gerald Supinski, Professor of Medicine, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Diaphragm EPA HMB
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Muscle Weakness
Keywords: diaphragm; limb muscle; EPA; HMB; ICU patients
MeSH Terms: conditions — Muscle Weakness | interventions — Docosahexaenoic Acids; Sodium Chloride; Fluoridation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control, to be given saline solution (Placebo Comparator): Intervention: This group will be given saline (30 ml every 12 hours) for 10 days
  Interventions: Drug: Saline
- EPA, eicosapentaenoic acid (Experimental): This group will be given 1000 mg EPA every 12 hours for 10 days
  Interventions: Drug: EPA, eicosapentaenoic acid
- HMB, hydroxymethylbutyrate (Experimental): This arm will be given HMB (1500 mg) every 12 hours for 10 days.
  Interventions: Drug: HMB, hydroxymethylbutyrate
- EPA and HMB (Experimental): Intervention: This group will be given EPA (1000 mg every 12 hours given via the GI tract) and HMB (1500 mg every 12 hours given via the GI tract) for 10 days.
  Interventions: Drug: HMB, hydroxymethylbutyrate; Drug: EPA, eicosapentaenoic acid

INTERVENTIONS:
Drug: HMB, hydroxymethylbutyrate — Hydroxymethylbutyrate will be given as 1500 mg powder dissolved in 30 ml saline given enterally every 12 hours for 7 days
  Other Names: This agent is an over the counter biopharmaceutical
  Arms: EPA and HMB; HMB, hydroxymethylbutyrate
Drug: EPA, eicosapentaenoic acid — EPA given as 1000 mg solution in saline (30 ml) administered enterally every 12 hours for 7 days
  Other Names: This is an over the counter biopharmaceutical
  Arms: EPA and HMB; EPA, eicosapentaenoic acid
Drug: Saline — Control
  Other Names: Salt water
  Arms: Control, to be given saline solution

SUMMARY:
The investigators will determine if administration of HMB (hydroxymethylbutyrate) or EPA (eicosapentaenoic acid) will increase diaphragm and limb muscle strength for patients on breathing machines in an intensive care unit. The investigators will first measure the strength of the diaphragm and a limb muscle (the quadriceps)using magnetic stimulators to activate these muscles. Muscle size will be measured by using an ultrasound to measure diaphragm thickness and quadriceps thickness. The investigators will also perform a vastus lateralis muscle biopsy. Patients will then be randomized to receive either placebo (saline 30 ml every 12 hours via the GI tract, EPA (1000 mg given every 12 hours via the GI tract), HMB (1500 mg given every 12 hours via the GI tract), or the combination of EPA (1000 mg given every 12 hours via the GI tract) and HMB (1500 mg given every 12 hours via the GI tract). Drugs will be given for 10 days; at the end of this time (on day 11), strength measurements, ultrasound muscle size measurements, and the vastus lateralis biopsy will be repeated. On day 21 an additional followup set of diaphragm and quadriceps strength and size measurements will be made (the biopsy will not be repeated for this last set of measurements). Patients will be followed clinically and patient outcomes (mortality, duration of mechanical ventilation after study entry) will be recorded.

DETAILED DESCRIPTION:
Objectives. There is a single objective for this study, namely, to determine if early administration of either EPA or HMB can prevent or reverse the development of respiratory muscle weakness in critically ill, mechanically ventilated patients. The investigators plan to randomize patients accepted into this protocol to administration of either a control (saline enteral control solution), EPA administration (enteral EPA), HMB (enteral HMB), or a combination of EPA and HMB. Drugs will be administered for 10 days and measurements of diaphragm and quadriceps strength and size will be performed immediately before (day 0) and immediately after (day 11) the period of drug administration. A third set of measurements (diaphragm and quadriceps strength and size) will be performed on day 21. Vastus lateralis muscle biopsies will also be taken on days 0 and 11; no biopsy will be performed for day 21 assessments. The investigators will also perform a chart review and assess ventilator mechanics (respiratory system static compliance and inspiratory airway resistance) at the time of the initial strength assessment. Patient outcomes (time on mechanical ventilation and mortality) will also be recorded. The investigators would expect that mean diaphragm strength and limb muscle strength measurements will be similar for four groups immediately before initiation of drug administration. The hypothesis will be supported if, post drug administration, diaphragm and limb muscle strength are higher for patients receiving EPA and/or HMB than the control group receiving no active drug.

Study Design.

The basic study design is to:

1. measure magnetic stimulated Pdi twitch and quadriceps strength and size, obtain a muscle biopsy from the vastus lateralis of the quadriceps, determine respiratory system compliance, determine airway resistance, and perform a chart review,
2. randomize patients to treatment with either: control solutions (30 ml of enteral saline solution every 12 hours), EPA (30 ml of enteral solution containing 1000 mg of EPA every 12 hours), HMB (30 ml of enteral solution containing 1500 mg HMB every 12 hours) or both EPA (30 ml of enteral solution containing 1000 mg of EPA every 12 hours) and HMB (30 ml of enteral solution containing 1500 mg HMB every 12 hours).
3. continue drugs for 10 days then
4. on day 11 remeasure magnetic stimulated Pdi twitch and quadriceps strength, repeat measurements of diaphragm and quadriceps size (i.e. thickness), repeat the vastus lateralis muscle biopsy, determine respiratory system compliance, determine airway resistance, and perform a chart review.
5. on day 21 remeasure magnetic stimulated Pdi twitch and quadriceps strength, and repeat measurements of diaphragm and quadriceps size (i.e. thickness), and perform another chart review.

For each chart review the investigators will obtain the following information: age, sex, diagnoses, reason for institution of mechanical ventilation, vital signs, bedside parameters of mechanical ventilation use (including mode of ventilation, duration of ventilation, level of oxygen, breath volume and rate, % triggered breaths), most recent arterial blood gas values, chest radiograph readings, recorded assessments of limb muscle strength and mental status.

Study Population. Adult patients requiring mechanical ventilation for more than 24 hours in one of the University of Kentucky adult ICU's will be asked to participate. Patients will be excluded if: (a) the physician caring for the patient determines that the patient is too unstable to tolerate these measurements, (b) if the patient requires high dose pressors (more than 15 mcg/min of norepinephrine or more than 15 mg/kg/min of dopamine), (c) if the patient requires more than 80% FiO2 or more than 15 cm H2O of PEEP, (d) if the patient has a cardiac pacemaker or implanted defibrillator, (e) if the patient has received neuromuscular blocking agents within the 48 hours preceding testing or has a known preexisting muscular disease, (f) if the patient has a recent history of variceal bleeding, and (g) if the patient is excessively sedated or mentally obtunded as judged by an inability to follow verbal commands. The investigators will also not study pregnant females, prisoners, or institutionalized decisionally impaired patients.

The goals are to recruit 80 patients into the study over a 24 month period (5 patients/month, 20 patients per experimental group). The investigators will study patients regardless of sex, race, or adult age. It is hoped that sufficient minorities and women will be studied so that the subject population is representative of the general patient population, but the investigators will be somewhat constrained by the numbers of available patients and the day to day makeup of the patient population in the UK ICU's. Inclusion of minorities and women will make the study results more generally applicable.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients requiring mechanical ventilation for more than 24 hours in one of the University of Kentucky adult ICU's

Exclusion Criteria:

* The physician caring for the patient determines that the patient is too unstable to tolerate these measurements,
* If the patient requires high dose pressors (more than 15 mcg/min of norepinephrine or more than 15 mg/kg/min of dopamine),
* If the patient requires more than 80% FiO2 or more than 15 cm H2O of PEEP,
* If the patient has a cardiac pacemaker or implanted defibrillator,
* If the patient has received neuromuscular blocking agents within the 48 hours preceding testing or has a known preexisting muscular disease,
* If the patient has a recent history of variceal bleeding,
* If the patient is excessively sedated or mentally obtunded as judged by an inability to follow verbal commands.
* We will not study pregnant females, prisoners, or institutionalized decisionally impaired patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2014-01; Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Supinski, MD, Principal Investigator — University of Kentucky
Locations (1):
- Chandler Hospital, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Supinski GS, Netzel PF, Westgate PM, Schroder EA, Wang L, Callahan LA. A randomized controlled trial to determine whether beta-hydroxy-beta-methylbutyrate and/or eicosapentaenoic acid improves diaphragm and quadriceps strength in critically Ill mechanically ventilated patients. Crit Care. 2021 Aug 26;25(1):308. doi: 10.1186/s13054-021-03737-9. PMID 34446067

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control, to be Given Saline Solution | EPA, Eicosapentaenoic Acid | HMB, Hydroxymethylbutyrate | EPA and HMB
Started | 20 | 17 | 18 | 18
Completed | 17 | 13 | 13 | 13
Not Completed | 3 | 4 | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control, to be Given Saline Solution | EPA, Eicosapentaenoic Acid | HMB, Hydroxymethylbutyrate | EPA and HMB | Total
Number analyzed (Participants) | 20 | 17 | 18 | 18 | 73
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 12 | 14 | 53
  >=65 years | 6 | 4 | 6 | 4 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58 [44 to 69] | 57 [40 to 65] | 64 [51 to 69] | 60 [46 to 64] | 59 [49 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 10 | 6 | 37
  Male | 10 | 6 | 8 | 12 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 2 | 12
  White | 18 | 13 | 14 | 15 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 17 | 18 | 18 | 73
Transdiaphragmatic pressure [Median (Inter-Quartile Range); unit: cm H2O] | 6 [4 to 9] | 4.7 [4 to 7] | 3.3 [2 to 4.7] | 6 [3 to 8] | 5 [3 to 7]

OUTCOME MEASURES:

1. Primary Outcome: Change of Skeletal Muscle Strength for One of the Drugs Compared to Placebo
Description: The primary outcome to be assessed is whether skeletal muscle strength (diaphragm and limb) has changed at the end of the administration trial (i.e. at 11 days) for patients given one or both of the active drugs (EPA or HMB) as compared to strength measurements at 11 days for patients given the placebo.
  The number of subjects in each group for this section represent the numbers for whom it was possible to measure trans-diaphragmatic pressure after completion of treatment regimens and thereby calculate a change in this parameter.
Time Frame: By the second strength measurement (11 days)
Population: Comparison of transdiaphragmatic twitch pressure (PdiTw), an index of strength, before and after treatment
Measure: Median (Inter-Quartile Range); unit: cm H2O
Arm/Group | Control, to be Given Saline Solution | EPA, Eicosapentaenoic Acid | HMB, Hydroxymethylbutyrate | EPA and HMB
Number analyzed (Participants) | 13 | 10 | 9 | 12
cm H2O | 1.3 [0 to 1.7] | 0.1 [-1.4 to 3.2] | 1.5 [0 to 3.2] | 0.7 [-1.8 to 3.7]

2. Secondary Outcome: Duration of Mechanical Ventilation
Description: Total duration on mechanical ventilation up to 50 days after study entry. The number of subjects in each group for this section represent the numbers for whom it was possible to determine the duration of mechanical ventilation after completion of treatment regimens.
Time Frame: Up to 50 Days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Control, to be Given Saline Solution | EPA, Eicosapentaenoic Acid | HMB, Hydroxymethylbutyrate | EPA and HMB
Number analyzed (Participants) | 13 | 10 | 9 | 12
Days | 5 [3 to 8] | 7 [7 to 13] | 6 [4.5 to 10] | 6 [3.8 to 7]

ADVERSE EVENTS:
Time Frame: Adverse event information was collected over the time the patient was in the study, i.e. the 10 days during which treatments were being given.
Description: Adverse events included all deaths and any unusual event during the time of study treatment. All adverse events were reported and reviewed by the University of Kentucky Clinical Translational Center Data Safety and Monitoring Board. The patients in this study were seriously ill, with a high predicted mortality. The deaths that occurred in this population were expected based on their clinical presentations, and all had failure of one or more organ systems.
Arm/Group | Control, to be Given Saline Solution | EPA, Eicosapentaenoic Acid | HMB, Hydroxymethylbutyrate | EPA and HMB
All-Cause Mortality (participants affected / at risk) | 0/20 | 2/17 | 1/18 | 2/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17 | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control, to be Given Saline Solution (N=20) | EPA, Eicosapentaenoic Acid (N=17) | HMB, Hydroxymethylbutyrate (N=18) | EPA and HMB (N=18)
Leg hematoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — One patient developed a leg hematoma two days after the initial set of measurements. This patient, however, also developed other limb hematomas several weeks after the study was over.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01270516/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01270516/SAP_001.pdf
  • Informed Consent Form (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT01270516/ICF_002.pdf